CLINICAL TRIAL: NCT00292968
Title: A Comprehensive Practice-Friendly Model for Promoting Healthy Behaviors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Collaborators: Robert Wood Johnson Foundation (Other); Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 6268
Record Dates: First submitted 2006-02-15; First posted 2006-02-16 (Estimated); Last update posted 2012-07-20 (Estimated); Status verified 2012-07

CONDITIONS: Unhealthy Diet, Exercise, Smoking, and Alcohol Use
Keywords: Health Behavior; Prevention; Informatics; Electronic Health Record
MeSH Terms: conditions — Motor Activity; Smoking; Alcohol Drinking; Health Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Computer based care
Behavioral: Telephone counseling
Behavioral: Group visits
Behavioral: Usual care

SUMMARY:
Using an electronic health record to link the resources of primary care practices and community programs will help patients to improve their diet and exercise, quit smoking, and moderate their drinking.

DETAILED DESCRIPTION:
We posit that practice systems to promote healthy behaviors must combine five attributes to be effective and sustainable. They must be comprehensive (addressing multiple behaviors and the "5 As"), flexible (offering options), generalizable to ordinary practices, practice-friendly (limiting burden), and apply the Chronic Care Model. We will test the effectiveness and implementation of an innovative "packaged" intervention with these features. Six ACORN-affiliated practices will adopt a brief (3 minute) routine to deliver A1-3 (Ask, Advise, Agree) in the office and to offer patients four options for intensive assistance (Assist [A4], Arrange [A5]) outside the office. Patients can select 9 months of online, telephone, or group counseling; or usual care. An electronic health record (EHR) will expedite the in-office intervention and referrals. Outcome measures will include health behaviors (derived from 7200 surveys administered pre-intervention and 3 and 9 months post-exposure) and implementation (derived from EHR data, "counselee" surveys, and patient/staff interviews). We hypothesize that implementing this novel "package" of interventions will be associated with improved health behaviors (using the Common Measures for physical activity, diet, smoking, and alcohol use). EHR-captured data will measure RE-AIM parameters, including Reach (14 sub-measures), Adoption, and Maintenance. Surveys and qualitative analysis of semi-structured interviews with patients and office staff will explore Implementation issues and suggested improvements. We hope to demonstrate that this innovative intervention not only promotes healthy behaviors but is feasible and sustainable in primary care. Accomplishing these goals requires a delicate balancing act--deploying evidence-based strategies that are effective in lifestyle change but limit demands for new staff, training, or time. We strike this balance by harnessing effective technologies and tools and by leveraging resources outside the practice. If our intervention helps patients change unhealthy behaviors and is appealing to ordinary practices, we envision the potential for widespread adoption and substantial population health benefits.

ELIGIBILITY:
Inclusion Criteria:

All individuals over the age of 8 years presenting for care in 9 primary care practices

Exclusion Criteria:

None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 5670 (Actual)
Dates: Start 2006-06; Primary Completion 2007-02 (Actual); Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Health behaviors (diet, exercise, smoking status, and alcohol use | 4 and 9 months post intervention

SECONDARY OUTCOMES:
Intervention's Reach, Adoption, Implementation, Maintenance | At the time of delivery of care

CONTACTS AND LOCATIONS:
Overall Officials: Alex Krist, MD, Study Director — Virginia Commonwealth University
Locations (1):
- Riverside Physicians Associates, Newport News, Virginia, United States

REFERENCES:
- [Background] Krist AH, Cifuentes M, Dodoo MS, Green LA. Measuring primary care expenses. J Am Board Fam Med. 2010 May-Jun;23(3):376-83. doi: 10.3122/jabfm.2010.03.090089. PMID 20453184
- [Result] Wilson DB, Johnson RE, Jones RM, Krist AH, Woolf SH, Flores SK. Patient weight counseling choices and outcomes following a primary care and community collaborative intervention. Patient Educ Couns. 2010 Jun;79(3):338-43. doi: 10.1016/j.pec.2010.01.025. Epub 2010 Mar 24. PMID 20338714
- [Result] Krist AH, Woolf SH, Johnson RE, Rothemich SF, Cunningham TD, Jones RM, Wilson DB, Devers KJ. Patient costs as a barrier to intensive health behavior counseling. Am J Prev Med. 2010 Mar;38(3):344-8. doi: 10.1016/j.amepre.2009.11.010. PMID 20171538
- [Result] Dodoo MS, Krist AH, Cifuentes M, Green LA. Start-up and incremental practice expenses for behavior change interventions in primary care. Am J Prev Med. 2008 Nov;35(5 Suppl):S423-30. doi: 10.1016/j.amepre.2008.08.007. PMID 18929990
- [Result] Krist AH, Woolf SH, Frazier CO, Johnson RE, Rothemich SF, Wilson DB, Devers KJ, Kerns JW. An electronic linkage system for health behavior counseling effect on delivery of the 5A's. Am J Prev Med. 2008 Nov;35(5 Suppl):S350-8. doi: 10.1016/j.amepre.2008.08.010. PMID 18929981
- See also: Source of funding - Prescription for Health Innitiative — http://www.prescriptionforhealth.org/
- See also: Practice base research network study conducting the study - ACORN — http://www.acorn.fap.vcu.edu/